CLINICAL TRIAL: NCT00242970
Title: Hypertrophic Scarring After Facial Burn: A Pilot, Observational Study of Static and Dynamic Measurements of Facial Scars With the 3-D Scanner Through the Scar Maturation Process
Brief Title: Hypertrophic Scarring After Facial Burn
Status: Completed | Type: Observational
Sponsor: Legacy Health System (Other)
Collaborators: Total Contact (Unknown)
Responsible Party: Principal Investigator, Helens Christians, Principal Investigator, Legacy Health System
Other Study IDs: OBC3DS-01
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: 3-Dimensional Color Scanning — Color imaging of the face and neck.
  Other Names: Cyberware 3030 RGB Color Scanner

SUMMARY:
Subjects with a burn to the face and/or neck will be enrolled into the study and a Three-Dimensional scanner used to see if it can objectively measure scar color and volume and measure the effect of scar on motion of the face and neck.

DETAILED DESCRIPTION:
Subjects will have 11 clinic visits over a 2-year period. An initial scan of the subject's head and neck will be made. Ten reproducible landmarks on the face and neck will be determined. The subject will return for follow up scans at Day 14, Day 28 and Month 2,6,9,12,18 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Face and/or Neck Burn

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes patients with burn injuries to their face and or neck.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Scar maturation | 5.5 years
  Can a 3-D scanner measure static and dynamic changes

CONTACTS AND LOCATIONS:
Overall Officials: Helen Christians, ORT/L, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Emanuel Hospital and Health Center, Portland, Oregon, United States